CLINICAL TRIAL: NCT05814068
Title: Active Screening of Arterial Hypertension by Community Outreach Workers in the Cayenne Metropolitan Area to Reduce the Incidence of Cardiovascular Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DEPIPREC
Record Dates: First submitted 2023-03-03; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-02

CONDITIONS: High Blood Pressure
Keywords: High blood pressure; Precarity; community outreach workers; Cardiovascular disease; Health care
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): diagnosis and treatment of high blood pressure
  Interventions: Drug: antihypertensive drug treatment

INTERVENTIONS:
Drug: antihypertensive drug treatment — Patients with hypertension will be treated for it by their physician

SUMMARY:
The main objective is to implement of a community-based primary care intervention against high blood pressure. We want to show that this intervention decreases the incidence of stroke in the community of agglomerations of the central coast of French Guiana, with a rapid effectiveness of about -30% at 2 years.

DETAILED DESCRIPTION:
The hypothesis of the research is that, thanks to a strategy of early detection of hypertension based on "outreach" by community relays, it will be possible to increase the effectiveness of primary prevention among the precarious population (early treatment, access to healthcare, improvement of therapeutic follow-up, reduction of renunciations and interruptions of treatment). This strategy, adapted to the Guianese context, would make it possible to reduce the incidence and mortality of cardiovascular diseases among the most vulnerable people, particularly stroke. Such data would be a prerequisite for a more ambitious strategy, aiming to implement policies on a sufficient scale policies on a scale and intensity sufficient to have an impact on the problem of social inequalities in health other than those related to high blood pressure.

The quasi-experimental before-and-after methodology makes it possible to compare, on a population basis, a quantitative endpoint - in this case the number of strokes - between before and after the implementation of a public health intervention. For reasons of acceptance by the partners, statistical power, and potential bias, a before-and-after design seems more interesting.

It will be a pre-screening of hypertension, a possible referral for medical care or opening of health care rights and health education through hygienic and dietary advice and health prevention focused on hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adults of at least 18 years old
* Residents of the agglomeration community of the central coast of French Guiana.

Exclusion Criteria:

* Person who has objected to participating in the study
* Person under guardianship or curatorship, persons under protective supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50000 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
To compare the incidence of stroke between before and after the start of the intervention according to PMSI data in resident persons in the agglomeration community of the central coast of French Guiana. | 5 years
  To compare the incidence of stroke between before and after the intervention

SECONDARY OUTCOMES:
The incidence of acute coronary syndrome (ACS), transient ischemic attack, lower extremity arterial disease, aneurysm and end stage renal disease treated. | comparison between before (over 5 years) and 1, 2 and 3 years after the beginning of the intervention according to PMSI data in the neighborhoods
Stroke incidence | comparison between before (over 5 years) and 1, 2 and 3 years after the beginning of the intervention according to PMSI data in the neighborhoods
treatment adherence | Inclusion
  lickert scale (5 levels)
Number of systolic and diastolic blood pressure measurements performed, number of new diagnoses and number of rediscoveries among those lost to follow-up during the intervention (number of people who give up on diagnosis or medical care) | 2 years
Quantification of the evolution of the prescription of antihypertensive drugs in Guiana via data from the Social Security | Before and 1, 2, and 3 years after the implementation of the intervention
stroke in hospital case fatality | 1, 2, and 3 years after the start of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu NACHER, PhD, Principal Investigator — Centre Hospitalier de Cayenne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mackenbach JP. Can we reduce health inequalities? An analysis of the English strategy (1997-2010). J Epidemiol Community Health. 2011 Jul;65(7):568-75. doi: 10.1136/jech.2010.128280. Epub 2011 Apr 1. PMID 21459930
- [Background] Mackenbach JP. Has the English strategy to reduce health inequalities failed? Soc Sci Med. 2010 Oct;71(7):1249-1253. doi: 10.1016/j.socscimed.2010.07.014. Epub 2010 Aug 3. No abstract available. PMID 20736133
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in hypertension prevalence and progress in treatment and control from 1990 to 2019: a pooled analysis of 1201 population-representative studies with 104 million participants. Lancet. 2021 Sep 11;398(10304):957-980. doi: 10.1016/S0140-6736(21)01330-1. Epub 2021 Aug 24. PMID 34450083
- [Background] Rochemont DR, Mimeau E, Misslin-Tritsch C, Papaix-Puech M, Delmas E, Bejot Y, DeToffol B, Fournel I, Nacher M. The epidemiology and management of stroke in French Guiana. BMC Neurol. 2020 Mar 24;20(1):109. doi: 10.1186/s12883-020-01650-2. PMID 32209060
- [Background] Rochemont DR, Lemenager P, Franck Y, Farhasmane A, Sabbah N, Nacher M. The epidemiology of acute coronary syndromes in French Guiana. Ann Cardiol Angeiol (Paris). 2021 Feb;70(1):7-12. doi: 10.1016/j.ancard.2020.09.032. Epub 2020 Oct 14. PMID 33067006
- [Background] Valmy L, Gontier B, Parriault MC, Van Melle A, Pavlovsky T, Basurko C, Grenier C, Douine M, Adenis A, Nacher M. Prevalence and predictive factors for renouncing medical care in poor populations of Cayenne, French Guiana. BMC Health Serv Res. 2016 Jan 28;16:34. doi: 10.1186/s12913-016-1284-y. PMID 26822003
- [Background] Van Melle A, Cropet C, Parriault MC, Adriouch L, Lamaison H, Sasson F, Duplan H, Richard JB, Nacher M. Renouncing care in French Guiana: the national health barometer survey. BMC Health Serv Res. 2019 Feb 6;19(1):99. doi: 10.1186/s12913-019-3895-6. PMID 30728033
- [Background] Hart JT. Commentary: Can health outputs of routine practice approach those of clinical trials? Int J Epidemiol. 2001 Dec;30(6):1263-7. doi: 10.1093/ije/30.6.1263. No abstract available. PMID 11821324
- [Background] Addo J, Ayerbe L, Mohan KM, Crichton S, Sheldenkar A, Chen R, Wolfe CD, McKevitt C. Socioeconomic status and stroke: an updated review. Stroke. 2012 Apr;43(4):1186-91. doi: 10.1161/STROKEAHA.111.639732. Epub 2012 Feb 23. PMID 22363052
- See also: Article - Bulletin épidémiologique hebdomadaire n.d — http://beh.santepubliquefrance.fr/beh/2020/2-3/2020_2-3_1.html
- See also: Rochemont DR, Dueymes JM, Roura R, Meddeb M, Couchoud C, Nacher M. End stage renal disease as a symptom of health inequalities in French Guiana. — http://doi.org/10.5114/jhi.2018.77646